CLINICAL TRIAL: NCT00639184
Title: Brain Research to Ameliorate Impaired Neurodevelopment (BRAIN): Home-based Intervention A Multicenter Trial of the Global Network for Women's and Children's Health Research
Brief Title: BRAIN - Home Intervention Trial
Acronym: BRAIN-HIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CP04; HD 40636
Record Dates: First submitted 2008-03-18; First posted 2008-03-20 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Asphyxia
Keywords: asphyxia; neurodevelopmental outcome; home counseling
MeSH Terms: conditions — Asphyxia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Home intervention program
  Interventions: Other: Early intervention counseling
- 2 (Active Comparator): health education counseling
  Interventions: Other: Health education counseling

INTERVENTIONS:
Other: Early intervention counseling — Bi-monthly home visits by counselor
  Arms: 1
Other: Health education counseling — World Health Education health education counseling program at home visits,twice per month
  Arms: 2

SUMMARY:
We plan to test a home-based parent-provided early developmental intervention (EI) both in infants with mild to moderate birth asphyxia and in infants without perinatal complications who will constitute a healthy comparison group in a randomized controlled trial. The trial will evaluate the effect of a resource-intensive early intervention (EI) program on the outcomes in infants born in rural communities in Zambia, India, and Pakistan. It will consist of frequent interaction (every 2 weeks the first year and every 4 weeks the second and third years) between parents and the parent trainer. The control group will receive enhanced health counseling (HC).

The overall goal will be to implement and evaluate an EI program for infants following birth asphyxia, which is sustainable in developing countries. The challenge will be to adapt programs demonstrated to be effective in developed countries to the circumstances of the developing world, while reducing the demands on resources. Because there are limited data on normative development and EI programs in developing countries, a group of infants without perinatal complications will also be randomized to the same conditions in order to provide a comparison of what may be achieved from the intervention in healthy infants in developing countries. A final aim will be to address individual variation in EI effects that could be due to child and/or family characteristics.

A randomized controlled experimental design will be used, in which infants who survive following birth asphyxia are randomly assigned to either EI or enhanced health education counseling (HC). The trial will randomize infants to a home-based parent-provided early developmental intervention (EI) with frequent home interaction between parents and parent trainers vs. HC. A group of infants without birth asphyxia or other major perinatal complications also will be randomized. Children will be examined by masked examiners at three time points (12, 24, and 36 month's assessments).

ELIGIBILITY:
Inclusion Criteria:

* birth asphyxia
* birth weight of at least 1,500g
* neurological examination consistent with normal, Stage I or II on the Ellis scale (Ellis, et al. 2000)
* willing to participate in an intervention program for 36 months.

Exclusion Criteria:

-

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
neurodevelopmental outcome | 36 months

SECONDARY OUTCOMES:
The improvements in cognitive, social, and motor development will be larger in the infants who have had birth asphyxia compared to those without birth asphyxia. | 12, 24 and 36 months
The effects of EI in infants with and without birth asphyxia will be moderated by child and family characteristics. | 12, 24 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Marion Koso-Thomas, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Wally A Carlo, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- JN Medical College, Belagavi, India
- Aga Khan University, Karachi, Pakistan
- University of Zambia, Lusaka, Zambia

REFERENCES:
- [Derived] Carlo WA, Goudar SS, Pasha O, Chomba E, McClure EM, Biasini FJ, Wallander JL, Thorsten V, Chakraborty H, Wright LL; Brain Research to Ameliorate Impaired Neurodevelopment-Home-based Intervention Trial Committee; National Institute of Child Health and Human Development Global Network for Women's and Children's Health Research. Neurodevelopmental outcomes in infants requiring resuscitation in developing countries. J Pediatr. 2012 May;160(5):781-5.e1. doi: 10.1016/j.jpeds.2011.10.007. Epub 2011 Nov 17. PMID 22099522
- [Derived] Wallander JL, McClure E, Biasini F, Goudar SS, Pasha O, Chomba E, Shearer D, Wright L, Thorsten V, Chakraborty H, Dhaded SM, Mahantshetti NS, Bellad RM, Abbasi Z, Carlo W; BRAIN-HIT Investigators. Brain research to ameliorate impaired neurodevelopment--home-based intervention trial (BRAIN-HIT). BMC Pediatr. 2010 Apr 30;10:27. doi: 10.1186/1471-2431-10-27. PMID 20433740